CLINICAL TRIAL: NCT04820764
Title: Early Feasibility Study of the CardioMech Mitral Valve Repair System (MVRS)
Brief Title: EFS of the CardioMech MVRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CardioMech AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 10228
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CardioMech Mitral Valve Repair System (MVRS) (Experimental)
  Interventions: Device: CardioMech MVRS

INTERVENTIONS:
Device: CardioMech MVRS — CardioMech MVRS

SUMMARY:
Safety and performance evaluation of the CardioMech Mitral Valve Repair System (MVRS) in patients with degenerative mitral valve regurgitation.

DETAILED DESCRIPTION:
The purpose of the clinical study is to obtain clinical data on the CardioMech Mitral Valve Repair System (MVRS) in patients diagnosed with moderate to severe (≥3+) or severe (≥4+), symptomatic, degenerative mitral regurgitation and who are determined to be at intermediate or high surgical risk for mitral valve repair, as assessed by the site's multidisciplinary heart team.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen (18) years of age or greater
* Moderate to severe (≥3+) or severe (≥4+) mitral valve regurgitation (per American Society of Echocardiography (ASE) guidelines) due to mitral valve prolapse or flail
* Intermediate or high surgical risk for mitral valve repair

Exclusion Criteria:

* History of rheumatic heart disease
* History of prior endocarditis
* History of prior repair or replacement of the mitral valve, or annuloplasty
* Severely calcified mitral leaflet or has evidence of calcification in the grasping area of the leaflets that would prevent leaflet anchor positioning and deployment
* Complex mechanism of MR (leaflet perforation, severe leaflet calcifications, commissural extension, commissural prolapse, multiple flail or prolapsing segments, cleft) present on required imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Freedom from serious adverse events determined to be related to the CardioMech MVRS device or procedure | 30 days
Change in MR grade | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Williams, MD, Principal Investigator — NYU Langone; Mayra Guerrero, MD, Principal Investigator — Mayo Clinic
Locations (12):
- United States (12):
  - Cardiovascular Institute of Los Robles Health System, Thousand Oaks, California
  - Northwestern University, Evanston, Illinois
  - Ascension St. Francis via Christi, Wichita, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - NYU Langone, New York, New York
  - Atrium Health Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ascension St. Thomas West, Nashville, Tennessee
  - Baylor Scott & White, The Heart Hospital, Plano, Texas
  - Intermountain Medical Center, Murray, Utah

IPD SHARING:
Plan to Share IPD: No